CLINICAL TRIAL: NCT02648607
Title: Management of Chronic Post-Partum Pelvic Girdle Pain Study: Evaluating Effectiveness of Combined Physiotherapy and a Dynamic Elastomeric Fabric Orthosis
Brief Title: Management of Chronic Post-Partum Pelvic Girdle Pain Study
Acronym: MOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Jenny Freeman, Professor in Physiotherapy and Rehabilitation, University of Plymouth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGP-LC15
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Pelvic Girdle Pain; Symphysis Pubis Dysfunction
Keywords: Pelvic Girdle Pain; Chronic Pelvic Girdle Pain; Symphysis Pubis Dysfunction; Sacroiliac Joint Dysfunction; Physiotherapy; Physical Therapy; Orthoses; Orthosis; Orthotic Devices
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Customised Orthosis (Experimental): Customised Dynamic Elastomeric Fabric Orthosis (DEFO)
  Interventions: Device: Customised Dynamic Elastomeric Fabric Orthosis (DEFO)

INTERVENTIONS:
Device: Customised Dynamic Elastomeric Fabric Orthosis (DEFO) — Eligible participants will be measured and fitted with a customised Dynamic Elastomeric Fabric Orthosis (DEFO). Participants will also be issued with standardised advice on PGP management via an information leaflet from Association of Chartered Physiotherapists in Women's health website.
  Other Names: Pelvic Support Garment; Customised Dynamic Elastomeric Fabric Orthosis

SUMMARY:
Pelvic Girdle Pain (PGP) during pregnancy occurs in approximately 70% of females and 38% of women continue to suffer PGP symptoms beyond 12 weeks following delivery. PGP post- partum causes pain during everyday activities that impacts negatively on health related quality of life and is associated with significant healthcare and societal costs. These women are often referred to physiotherapy, however management is difficult and there is a weak evidence base for its management.

Alongside the provision of advice and information, physiotherapists commonly prescribe orthoses such as a rigid belt with the aim of optimising pelvic stability and reducing pain. More recently a novel customised Dynamic Elastomeric Fabric Orthosis has been developed as an alternative to an 'off the shelf' pelvic belt. No studies have investigated their effectiveness in complementing standard physiotherapy advice and management.

The investigators will undertake a comprehensive systematic review of the literature to critically evaluate the evidence base for the conservative management of chronic post-partum PGP. This will inform a single case experimental design. Here eight AB single case studies will be performed with the point of intervention being randomised between subjects. The use of a randomisation test permits subsequent statistical analyses of group effects. Participants' pain, activity levels, and quality of life will be evaluated along with subjective changes in confidence and urinary incontinence. Adherence to orthosis use will be diarised. Exit interviews will assess aspects such as the appropriateness of the outcome measures and acceptability of the intervention that will help to inform future clinical trials.

DETAILED DESCRIPTION:
Pelvic girdle pain (PGP) occurs in 70% of pregnant women; of whom 25% have severe pain and 8% severe disability requiring the use of crutches, wheelchair or confinement to bed (Wu et al, 2004). At a personal level, women with PGP find that everyday activities such as turning in bed, prolonged walking, or carrying items may cause pain; impacting negatively on quality of life (Wang et al, 2004). In economic terms societal costs are significant, mainly as a consequence of work absenteeism; with 20% of people requiring an average of 7 weeks sick leave (Noren et al, 1997). The impact of this problem is significant; with 812, 970 deliveries occurring throughout the UK in 2012/13 (http://www.statistics.gov.uk/hub/index.html). Pregnancy related PGP has also been documented to increase.

PGP during pregnancy is thought to occur due to increased pelvic joint motion as a consequence of hormonal and biomechanical factors. For many women PGP symptoms resolve within approximately 3 months of delivery, however, approximately 38% of females continue to experience pain beyond 3 months following delivery (Gutke et al 2010, Van de Pol et al 2006). It is unknown why chronic symptoms persist, but age, parity, pre- pregnancy body mass index (BMI), mode of delivery and previous PGP, along with emotional and psychosocial factors have been identified as risk factors associated with chronic PGP (Robinson et al, 2010)). Further, women having caesarean section are at increased risk of post-partum chronic PGP, which is noteworthy given the increasing percentage of women who are electing for caesarean section for early symptomatic relief of peri-partum PGP. Urinary incontinence is also documented to affect approximately 70% of females suffering with pregnancy related PGP. If PGP symptoms continue into the post-partum then urinary incontinence is reported to continue due to an association with PGP and pelvic floor muscle weakness (Fitzgerald et al, 2012).

PGP is difficult to manage with limited guidance from the literature on conservative management. European Guidelines recommend exercise prescription for PGP (Vleeming et al., 2008) leading to the development of a Specialist Women's Health group information booklet that will be used in the current study.

An integral part of physiotherapists' management approach for PGP is the provision of orthoses such as rigid pelvic belts, which aim to improve pelvic joint stability and thus reduce pain. Pelvic belts apply forces to the pelvis within the transverse plane. Recently dynamic elastomeric fabric orthoses (DEFO) have been developed. A DEFO is made of elastomeric panels (e.g. Lycra ®) that are pre-stretched and can provide forces in multiple directions to the pelvis. Thus they provide continued multi-axis support whilst being flexible enough to allow people to participate in everyday activities. Studies on sports people with pelvic girdle pain have shown that the application of forces in more than one plane decreases pain and improves function over and above that seen with the application of transverse forces associated with pelvic belts (Sawle et al, 2013). Therefore the DEFO may have advantages over current rigid pelvic belts in terms of mode of action, clinical effectiveness and user satisfaction. To date a comprehensive literature search has revealed there have been no trials of orthotic use in women with chronic PGP post-partum. This project will therefore follow the recommendations of the Medical Research Council in the development and evaluation of complex interventions to establish a clearer understanding of PGP and its management post-partum that can inform future clinical trials.

ELIGIBILITY:
Inclusion Criteria: Women with PGP (commenced or aggravated during pregnancy) will be included if they:

* have symptoms that continued for > 3 months following birth,
* have PGP that causes walking and/or stair climbing to be bothersome (as determined by a score of at least 2 on a 10 point visual analogue scale)
* are positive on at least 3 out of 7 pain provocation tests (see screening section below)

Exclusion Criteria: Women will be excluded if they have:

* A recent history/signs or symptoms indicative of serious causes of pain that might be inflammatory infective, traumatic, neoplastic, degenerative or metabolic.

In particular exclusion will occur if following questioning or clinical examination there is evidence of:

* trauma
* Indicators of serious pathology
* steroid use
* drug abuse
* HIV infection
* immunosuppressed state
* neurological symptoms/signs (including cauda-equina)
* fever
* systemically unwell
* obstetric complications
* pain that does not improve with rest/severe disabling pain
* history of chronic back or pelvic pain requiring surgery.
* a known skin allergy to Lycra

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Pain Levels | Baseline (Pre intervention), 1 weekly intervals for 8, 9, 10 weeks (dependent on baseline randomisation), then a following 8,9,10 weeks Intervention (total 16 weeks)
  Change in pain levels at 1 weekly intervals will be measured by a self-report numerical pain rating scale

SECONDARY OUTCOMES:
Activity Levels | Baseline (Pre intervention), 1 weekly intervals for 8, 9, 10 weeks (dependent on baseline randomisation), then a following 8,9,10 weeks Intervention (total 16 weeks)
  Change in activity levels at 1 weekly intervals will be measured by a self-report questionnaire
Quality if Life | Baseline (Pre intervention), 1 weekly intervals for 8, 9, 10 weeks (dependent on baseline randomisation), then a following 8,9,10 weeks Intervention (total 16 weeks)
  Change in quality of life levels at 1 weekly intervals will be measured by a self-report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lee Cameron, Principal Investigator — University of Plymouth
Locations (2):
- United Kingdom (2):
  - Southmead Hospital, Bristol, Avon
  - University of Plymouth, Plymouth, Devon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu WH, Meijer OG, Uegaki K, Mens JM, van Dieen JH, Wuisman PI, Ostgaard HC. Pregnancy-related pelvic girdle pain (PPP), I: Terminology, clinical presentation, and prevalence. Eur Spine J. 2004 Nov;13(7):575-89. doi: 10.1007/s00586-003-0615-y. Epub 2004 Aug 27. PMID 15338362
- [Background] Wang SM, Dezinno P, Maranets I, Berman MR, Caldwell-Andrews AA, Kain ZN. Low back pain during pregnancy: prevalence, risk factors, and outcomes. Obstet Gynecol. 2004 Jul;104(1):65-70. doi: 10.1097/01.AOG.0000129403.54061.0e. PMID 15229002
- [Background] Noren L, Ostgaard S, Nielsen TF, Ostgaard HC. Reduction of sick leave for lumbar back and posterior pelvic pain in pregnancy. Spine (Phila Pa 1976). 1997 Sep 15;22(18):2157-60. doi: 10.1097/00007632-199709150-00013. PMID 9322326
- [Background] Gutke A, Sjodahl J, Oberg B. Specific muscle stabilizing as home exercises for persistent pelvic girdle pain after pregnancy: a randomized, controlled clinical trial. J Rehabil Med. 2010 Nov;42(10):929-35. doi: 10.2340/16501977-0615. PMID 21031289
- [Background] van de Pol G, de Leeuw JR, van Brummen HJ, Bruinse HW, Heintz AP, van der Vaart CH. The Pregnancy Mobility Index: a mobility scale during and after pregnancy. Acta Obstet Gynecol Scand. 2006;85(7):786-91. doi: 10.1080/00016340500456373. PMID 16817074
- [Background] Robinson HS, Mengshoel AM, Veierod MB, Vollestad N. Pelvic girdle pain: potential risk factors in pregnancy in relation to disability and pain intensity three months postpartum. Man Ther. 2010 Dec;15(6):522-8. doi: 10.1016/j.math.2010.05.007. PMID 20621546
- [Background] Fitzgerald CM, Santos LR, Mallinson T. The association between pelvic girdle pain and urinary incontinence among pregnant women in the second trimester. Int J Gynaecol Obstet. 2012 Jun;117(3):248-50. doi: 10.1016/j.ijgo.2012.01.014. Epub 2012 Mar 28. PMID 22459920
- [Background] Vleeming A, Albert HB, Ostgaard HC, Sturesson B, Stuge B. European guidelines for the diagnosis and treatment of pelvic girdle pain. Eur Spine J. 2008 Jun;17(6):794-819. doi: 10.1007/s00586-008-0602-4. Epub 2008 Feb 8. PMID 18259783
- [Background] Sawle L, Freeman J, Marsden J, Matthews MJ. Exploring the effect of pelvic belt configurations upon athletic lumbopelvic pain. Prosthet Orthot Int. 2013 Apr;37(2):124-31. doi: 10.1177/0309364612448806. Epub 2012 Jul 2. PMID 22751218